CLINICAL TRIAL: NCT06310044
Title: Evaluation of Commiphora Myrrh Versus Sodium Hypochlorite as Root Canal Irrigant on Post- Operative Pain and Bacterial Load Reduction in Symptomatic Mandibular Premolar Teeth With Necrotic Pulp. (A Randomized Clinical Trial)
Brief Title: Effect of Commiphora Myrrh Solution as a Root Canal Irrigant on Post Operative Pain and Bacterial Load Reduction in Necrotic Tooth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rahaf Abdullah khalel manzalawi, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Commiphora Myrrh
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Necrotic Pulp
Keywords: Asymptomatic Necrotic Mandibular Premolar
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commiphora Myrrh (Experimental): 50% Commiphora Myrrh
  Interventions: Other: Root canal irrigant Commiphora Myrrh 50%
- Sodium hypochlorite (Active Comparator): 2.5% NaOCl
  Interventions: Other: Root canal irrigant Commiphora Myrrh 50%

INTERVENTIONS:
Other: Root canal irrigant Commiphora Myrrh 50% — Root canal irrigant

SUMMARY:
Clinically compare the post-operative pain , incidences post-operative swelling , post-operative number of analgesic tablets taken by patient and amount of bacterial load reduction after using 50% Commiphora Myrrh Chemomechanical preparation , versus 2.5% NaOCl,in asymptomatic necrotic mandibular premolar treated in single visit.

DETAILED DESCRIPTION:
The patients will be randomly divided into 2 groups. Intervention group (50% Commiphora Myrrh solution root canal irrigant) and control group (2.5% sodium hypochlorite root canal irrigant)

Post-operative pain will be measured at 6,12,24,48 hours post-operatively The pain will be recorded using numerical rating scale

Post-operative swelling will be measured at 6,12,24,48 hours post-operatively The swelling will be receded using visual swelling rating scale

Number of analgesic tablets taken by the patient post-operatively. Up to 48 hours

Amount of bacteria load reduction The intracanal bacterial load reduction will be determined using agar culture technique by counting the colony forming units per milliliter (CFI /ml) before and after root canal preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patient (ASA I, II).
2. Age between 20 and 40 years.
3. Male or female.
4. Patient who is able to sign and comprehend the pain scale (committed patient).
5. Mandibular single rooted premolars having the following criteria:

   * With single root canal.
   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pulpal pain.
   * Positive pain on percussion denoting apical periodontitis.
   * Slight widening of periodontal space or peri-apical radiolucency smaller than 3 mm (0-2mm)

Exclusion Criteria:

1. Medically compromised patients (ASA III or IV).
2. Teeth with:
3. Patients who could not interpret the NRS.

   * Immature roots.
   * Vital pulp tissues.
   * Association with swelling.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III.
   * Previously accessed or endodontically treated.
   * Deep periodontal pockets more than 4 mm.
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
4. Patients with diabetes, immune-compromising, and immunosuppression disease and pregnant women will be also excluded.
5. History of intolerance to NSAIDs.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | Post-operative pain measured at 6,12,24,48 hours after single visit Treatment
  Categorical None 0 Mild 1-3 Moderate 4-6 Sever 7-10

SECONDARY OUTCOMES:
incidence of Post-operative swelling | Up to 48 hours post-
  Categorical Of visual swelling scale of post- operative

OTHER OUTCOMES:
Amount of intracanal Bacterial CFUs/ml | Pre-intervention, pre-instrumentation after access cavity. Post-instrumentation up to 10min
  Intra canal bacterial load reduction will be determined using agar culture technique by counting the colony forming units per milliliter (CFUs/ml) before and after root canal preparation
Number of analgesic Counting Tablets taken by the patient after endodontic treatment | Up to 48hours post-operative
  Counting the tablet after the treatment

IPD SHARING:
Plan to Share IPD: Yes